CLINICAL TRIAL: NCT03793244
Title: The Augmented Versus Routine Approach to Giving Energy Trial Metabolic Effects Sub-study (TARGET-ME)
Brief Title: TARGET-Metabolic Effects
Acronym: TARGET-ME
Status: Completed | Type: Observational
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Collaborators: The Canberra Hospital (Other); Royal Adelaide Hospital (Other); Auckland City Hospital (Other Government); Melbourne Health (Other)
Responsible Party: Principal Investigator, anzicrc, ICU Nutrition Research Program Manager, Australian and New Zealand Intensive Care Research Centre
Other Study IDs: MC_001 V1 240217
Record Dates: First submitted 2017-04-23; First posted 2019-01-04 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Critical Illness; Enteral Nutrition
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental: TARGET protocol EN 1.5 kcal/mL: Enteral (EN) feed 1.5 kcal/mL. Indirect calorimetry and/or VCO2 measurements will be taken periodically while in the TARGET main study
  Interventions: Dietary Supplement: TARGET protocol EN 1.5 kcal/mL
- Active Comparator: TARGET protocol EN 1.0 kcal/mL: Enteral feed 1.0 kcal/mL Indirect calorimetry and/or VCO2 measurements will be taken periodically while in the TARGET main study

INTERVENTIONS:
Dietary Supplement: TARGET protocol EN 1.5 kcal/mL — Enteral nutrition
  Groups: Experimental: TARGET protocol EN 1.5 kcal/mL

SUMMARY:
The estimation of calorie needs during routine practice in critically ill patients is highly variable and the thermogenic effect of continuous delivery of enteral nutrition (EN) on overall calorie utilisation in critically ill adults is unknown. The TARGET-ME study is a substudy of the TARGET trial (NCT02306746). The TARGET trial provides the perfect opportunity to measure calorie utilisation via indirect calorimetry (IC) and ventilator-derived carbon dioxide production (VCO2) to compare measured calorie utilisation to estimation methods, determine the potential thermic effect of EN solutions with different energy concentrations and investigate any associations with outcome.

ELIGIBILITY:
Inclusion Criteria:

Patients must first meet the inclusion and none of the exclusion criteria for the TARGET main trail (NCT02306746). The following additional criteria applies for this study when indirect calorimetry is being used:

* Within 48 hours of randomisation to TARGET (first measurement only)
* Fi02 < 50% for the past 1 hour
* Positive end expiratory pressure (PEEP) < 12 mmHg for the past 1 hour
* The IC test can be conducted within 48 hours of randomisation to TARGET
* The patient is not considered agitated using the usual site assessment
* There is a clinician available to complete the test

Exclusion Criteria:

* There is an air leak in the ventilation circuit (ie bubbling inter-costal catheters, cuff leak at the endotracheal tube
* The patient is receiving renal replacement therapy or extracorporeal membrane oxygenation at the time of measurement
* Has had surgery in the last 6 hours (if enough time within the 48 hour window, consider waiting until this criteria is less than 6 hours)
* If the patient has a traumatic brain injury, for the previous 6 hours, their intracranial pressures have been unstable and in the opinion of the treating intensivist are not controlled
* The treating clinician believes that the IC test will pose risk to the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult critically ill patients who are mechanically ventilated
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Calorie difference in kcal | Up to day 28
  Difference in mean calorie delivery and mean measured calorie utilisation over the study period (expressed as a percentage of measured requirements received) in each study group

SECONDARY OUTCOMES:
Calorie difference in kcal in the whole study cohort | Up to day 28
  Calorie difference in kcal between mean calorie delivery and mean measured calorie utilisation over the study period (expressed as a percentage of measured requirements received) in the whole study cohort

OTHER OUTCOMES:
Calorie difference in kcal | Up to day 28
  Calorie difference in kcal between mean measured calorie utilisation and mean calorie requirements predicted by the estimation method used in TARGET and in routine clinical practice
Energy balance | Up to day 28
  Energy balance in both the intervention and standard care groups (with measured calorie utilisation as the reference) up until 4 weeks post randomisation
Degree of diet induced thermogenesis | Up to day 28
  measured as the difference between mean measured calorie utilisation in kcal between the two intervention groups
Correlation of energy expenditure (EE) assessed by IC and VCO2 compared to predictive equations estimates of EE | Up to day 28
  Correlation (bias, precision, accuracy rates) of EE assessed by IC and VCO2 compared to predictive equations estimates of EE

CONTACTS AND LOCATIONS:
Locations (1):
- ANZIC-RC, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No